CLINICAL TRIAL: NCT05249400
Title: Effect of Off-site Assistance on Success Rate of Selective Cannulation During Hands-on ERCP Training: A Randomized Non-inferiority Trial
Brief Title: Effect of Off-site Assistance on Success Rate of Selective Cannulation During hands-on ERCP Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20201005-2
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: ERCP Training; Biliary Tract Diseases; Pancreatic Diseases
MeSH Terms: conditions — Biliary Tract Diseases; Pancreatic Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Off-site assistance group (Experimental): The trainer supervised the trainee's cannulation operation outside the procedure room through a high-definition screen displaying the endoscopic and fluoroscopic view. The trainer was allowed to provide unlimited verbal instructions to the trainee by an intercom. The trainer was not allowed to enter the procedure room and touch the endoscope or accessories until the trainee ask for help or failed to achieve deep biliary cannulation. The trainer would halt and correct the trainee's inappropriate maneuvers immediately to avoid unnecessary papillary trauma and potential complications. Then the trainer would then take over and continue with the cannulation.
  Interventions: Procedure: Off-site assistance
- On-site assistance group (No Intervention): The trainer supervised the trainee's cannulation operation in the procedure room. The trainer was allowed to provide unlimited verbal instructions to the trainee on-site. The trainer was not allowed to touch the endoscope or accessories until the trainee ask for help or failed to achieve deep biliary cannulation. The trainer would halt and correct the trainee's inappropriate maneuvers immediately to avoid unnecessary papillary trauma and potential complications. Then the trainer would then take over and continue with the cannulation.

INTERVENTIONS:
Procedure: Off-site assistance — The trainer supervised the trainee's cannulation operation outside the procedure room through a high-definition screen displaying the endoscopic and fluoroscopic view. The trainer was allowed to provide unlimited verbal instructions to the trainee by an intercom.
  Arms: Off-site assistance group

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is a technically challenging procedure. It takes time to learn the basic skills and need at least 180 - 200 cases for trainees to achieve competency in ERCP. Hands-on practice in patients remains the gold standard for ERCP training. Traditional hands-on ERCP training requires the trainer to be on-site to assist the trainee with ERCP operations. We hypothesized that the trainee can be safely guided by trainer off-site with interactive audio and endoscopic and fluoroscopic view. Technology-enabled health care at a distance has profound scientific potential and accordingly has been met with growing interest. Teleguidance facilitated ERCP cannulation is a strategy to provide expert cannulation guidance to trainee in settings where such expertise is not on-site. Teleguidance not only reduces unnecessary radiation exposure of endoscopist, but also provides remote assistance for trainees to complete training or further improve skills. Given the advantages of the off-site teleguidance, it could be an attractive substitute for on-site hands-on ERCP training.

The primary aim of this study was to evaluate whether off-site assistance (Off group) could achieve a comparable success rate to on-site assistance (On group) regarding the rates of successful selective biliary cannulation during ERCP training.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years old
* With native papilla

Exclusion Criteria:

* History of partial or total gastrectomy (Billroth I/II, Roux-en-Y)
* Type II duodenal stenosis
* Previously failed cannulation
* Chronic pancreatitis with stones in the pancreatic head
* Hemodynamic instability
* Lactating or pregnant women
* Inability to give written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of selective cannulation by trainee | up to one year
  The rate of successful selective cannulation by trainee during the training period.

SECONDARY OUTCOMES:
Complication rate | up to one year
  Post-ERCP pancreatitis (mild, moderate-to-severe); Hyperamylasemia; Cholangitis (mild, moderate, severe); Perforation (conservative therapy, surgery）; Bleeding (mild, moderate, severe);
Performance score of selective cannulation | up to one year
  The trainee's performance score of cannulation by trainer and performance video. Out of 5 points, higher scores are better
Final success rate of cannulation | up to one year
  The overall rate of successful selective cannulation by trainee and trainer
Total time of successful cannulation | up to one year
  Total time required for successful cannulation
Radiation exposure time | up to one year
  Radiation exposure time for trainee and trainer

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Pan Y, Zhao L, Leung J, Zhang R, Luo H, Wang X, Liu Z, Wan B, Tao Q, Yao S, Hui N, Fan D, Wu K, Guo X. Appropriate time for selective biliary cannulation by trainees during ERCP--a randomized trial. Endoscopy. 2015 Aug;47(8):688-95. doi: 10.1055/s-0034-1391564. Epub 2015 Mar 6. PMID 25750038
- [Background] Wani S, Han S, Simon V, Hall M, Early D, Aagaard E, Abidi WM, Banerjee S, Baron TH, Bartel M, Bowman E, Brauer BC, Buscaglia JM, Carlin L, Chak A, Chatrath H, Choudhary A, Confer B, Cote GA, Das KK, DiMaio CJ, Dries AM, Edmundowicz SA, El Chafic AH, El Hajj I, Ellert S, Ferreira J, Gamboa A, Gan IS, Gangarosa L, Gannavarapu B, Gordon SR, Guda NM, Hammad HT, Harris C, Jalaj S, Jowell P, Kenshil S, Klapman J, Kochman ML, Komanduri S, Lang G, Lee LS, Loren DE, Lukens FJ, Mullady D, Muthusamy RV, Nett AS, Olyaee MS, Pakseresht K, Perera P, Pfau P, Piraka C, Poneros JM, Rastogi A, Razzak A, Riff B, Saligram S, Scheiman JM, Schuster I, Shah RJ, Sharma R, Spaete JP, Singh A, Sohail M, Sreenarasimhaiah J, Stevens T, Tabibian JH, Tzimas D, Uppal DS, Urayama S, Vitterbo D, Wang AY, Wassef W, Yachimski P, Zepeda-Gomez S, Zuchelli T, Keswani RN. Setting minimum standards for training in EUS and ERCP: results from a prospective multicenter study evaluating learning curves and competence among advanced endoscopy trainees. Gastrointest Endosc. 2019 Jun;89(6):1160-1168.e9. doi: 10.1016/j.gie.2019.01.030. Epub 2019 Feb 7. PMID 30738985
- [Background] Pahlsson HI, Groth K, Permert J, Swahn F, Lohr M, Enochsson L, Lundell L, Arnelo U. Telemedicine: an important aid to perform high-quality endoscopic retrograde cholangiopancreatography in low-volume centers. Endoscopy. 2013;45(5):357-61. doi: 10.1055/s-0032-1326269. Epub 2013 Mar 6. PMID 23468194
- [Background] Brinne Roos J, Bergenzaun P, Groth K, Lundell L, Arnelo U. Telepresence-teleguidance to facilitate training and quality assurance in ERCP: a health economic modeling approach. Endosc Int Open. 2020 Mar;8(3):E326-E337. doi: 10.1055/a-1068-9153. Epub 2020 Feb 21. PMID 32118106
- [Background] Shimizu S, Itaba S, Yada S, Takahata S, Nakashima N, Okamura K, Rerknimitr R, Akaraviputh T, Lu X, Tanaka M. Significance of telemedicine for video image transmission of endoscopic retrograde cholangiopancreatography and endoscopic ultrasonography procedures. J Hepatobiliary Pancreat Sci. 2011 May;18(3):366-74. doi: 10.1007/s00534-010-0351-8. PMID 21127912